CLINICAL TRIAL: NCT01678469
Title: Lipophilic Micronutrients, Adipokines and Gestational Diabetes Mellitus
Acronym: 2011-23
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-A001138-33
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational | interventions — Blood Specimen Collection

ARMS (1):
- blood sample (Other)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
Background Gestational diabetes mellitus (GDM) is defined as a defect of glucose tolerance with its onset or its first recognition during pregnancy and that usually disappears, at least temporarily, after delivery. Its prevalence generally ranges between 3 and 6%, but may reach 12 to 15% in high-risk populations or specific ethnic groups. GDM increases the risk of potentially severe maternal, fetal and neonatal complications (gestational hypertension, pre-eclampsia, caesarean delivery; macrosomia; shoulder dystocia). These risks are linearly correlated with the level of maternal hyperglycaemia. GDM is due to a failure of pancreatic beta cells to sustain compensatory insulin secretion for insulin resistance that is physiological in pregnancy but can be much more pronounced in some women, especially in case of overweight or obesity. Maternal obesity is a major risk factor of GDM. Yet, micronutrient deficiencies are frequently reported in obese patients. Some nutritional deficiencies, concerning particularly some lipophilic micronutrients (vitamin A, vitamin D, vitamin E, carotenoids) may be associated with diseases linked to insulin resistance. Numerous studies show an inverse relationship between plasma concentrations and/or dietary intake of these micronutrients and incidence of type 2 diabetes. Vitamin D deficiency could be involved in the pathogenesis of type 2 diabetes through an alteration of insulin secretion and sensitivity. Deficiencies in vitamin A, vitamin E or carotenoids (in particular lycopene and beta carotene) increase oxidative stress and pro-inflammatory status, and could thus be implied in the physiopathology of insulin resistance and glucose intolerance.

Some case-control studies find an inverse correlation between the plasma concentrations of vitamin D during pregnancy and the incidence of GDM, independently of age, ethnic origin and of body mass index. Data are scarce for vitamin A and vitamin E, and are lacking for carotenoids. Besides, the few available studies are mainly descriptive ones, without clear explanations on underlying mechanisms. The favourable effects of these micronutrients on insulin sensitivity could be partially mediated by adipokines and/or pro-inflammatory cytokines secreted at the level of the adipose tissue. Numerous studies showed that women developing GDM during their pregnancy presented with a significant decrease in the circulating rates of adiponectin, (that is an adipokine with anti-inflammatory and insulin-sensitizing properties) and a significant increase in the secretion of the pro-inflammatory cytokines implied in the physiopathology of insulin resistance. In our laboratory (INRA unit 1260), we showed in experimental works conducted in vitro in human adipocytes and in vivo in mice that vitamin E could induce the transcription and the secretion of adiponectin; we also showed that vitamin D or lycopene could modulate the inflammatory reaction in the adipose tissue, which is involved in the physiopathology of insulin resistance.

Aims and methods We hypothesise that, in pregnant women, there is a link between plasma concentrations and dietary intakes of lipophilic micronutrients (mainly vitamins A, D, E and carotenoids), secretion of adipokines and pro-inflammatory cytokines, and risk of developing a GDM; we also hypothesise that this relationship is independent of age, body mass index, ethnic origin and other main risk factors of GDM. To test this hypothesis, we aim to lead a transversal monocentric study, within a population of 500 pregnant women submitted to a systematic screening of GDM by an oral glucose tolerance test (OGTT) in the Hôpital Nord of Marseilles.

The main criterion of evaluation of the link between lipophilic micronutrients and GDM will be a nutritional score calculated as follows: for each micronutrient (vitamin A, D, E, lycopene, beta carotene, alpha carotene, lutein), we will attribute 0 point if the patient is situated in the lowest quartile, 1 or 2 points in the following quartiles, and 3 points in the highest quartile. At the end, each patient will thus have a score between 0 and 21 reflecting the global status of these micronutrients.

The main secondary objectives will be to define the relationships between the plasma concentrations and dietary intakes of these micronutrients and 1/the value of glycemia and insulinemia during OGTT 2/the degree of insulin sensitivity estimated by the measure of HOMA index, 3/the circulating rates of some adipokines (mainly adiponectin, leptin, chemerin) and pro-inflammatory cytokines (TNF alpha, IL-1, IL-6), and 4/the children's birth weight.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman screen for Gestational diabetes mellitus (GDM)

Exclusion Criteria:

* pregnant woman with intercurate disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2015-01-21 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
link between plasma concentrations and dietary intakes of lipophilic micronutrients and risk of developing a Gestational diabetes mellitus | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assitance Publique Hôpitaux de Marseille, Marseille, France